CLINICAL TRIAL: NCT02072980
Title: Evaluation of the Lubricity of DAILIES TOTAL1® Contact Lenses After Wear
Brief Title: DAILIES TOTAL1® Lubricity Post Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: M-14-002
Record Dates: First submitted 2014-02-24; First posted 2014-02-27 (Estimated); Results first posted 2015-05-14 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-04

CONDITIONS: Refractive Error
Keywords: DT1; DAILIES TOTAL1®; Lubricity
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 16hrs/15mins (Other): Delefilcon A contact lenses worn bilaterally (in both eyes) for 16 waking hours (1 day) in Period 1, followed by 15 minutes in Period 2. A fresh pair of lenses was dispensed for Period 2.
  Interventions: Device: Delefilcon A contact lenses
- 15mins/16hrs (Other): Delefilcon A contact lenses worn bilaterally for 15 minutes in Period 1, followed by 16 waking hours (1 day) in Period 2. A fresh pair of lenses was dispensed for Period 2.
  Interventions: Device: Delefilcon A contact lenses

INTERVENTIONS:
Device: Delefilcon A contact lenses — Silicone hydrogel contact lenses
  Other Names: DAILIES TOTAL1®

SUMMARY:
The primary objective of the study is to demonstrate that the lubricity of DAILIES TOTAL1® (DT1) lenses after 16 hours of wear is equivalent to the lubricity of unworn DT1 lenses.

DETAILED DESCRIPTION:
In this study, participants wore study lenses for 2 specified time periods (16 hours and 15 minutes, treatment sequence randomized) following which lenses were collected for ex vivo lubricity analysis. The ex vivo lubricity analysis was evaluated under a separate non-clinical protocol.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign Informed Consent document.
* Adapted, current soft contact lens wearer.
* Requires contact lens powers within the specified range of -0.50 diopters (D) to -10.00D.
* Cylinder between 0.00D and -1.00D (inclusive) in both eyes at Visit 1 manifest refraction.
* Vision correctable to 20/25 or better in each eye at distance with study lenses.
* Willing to wear study lenses at least 16 waking hours in one day and attend all study visits.
* Able to be successfully fitted with study lenses.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Any ocular infection, inflammation, abnormality or active disease that would contraindicate contact lens wear, as determined by the Investigator.
* Use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the Investigator.
* Use of artificial tears and rewetting drops during the study.
* Monocular (only one eye with functional vision) or fit with only one lens.
* Any abnormal ocular condition observed during the Visit 1 slit lamp examination.
* History of herpetic keratitis, ocular surgery, or irregular cornea.
* Pregnant.
* Participation in any clinical study within 30 days of Visit 1.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa L. Zoota, MPH, CCRA, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1 study center located in the US.
Pre-assignment Details: This reporting group includes all randomized participants (15).
Groups:
- 16hr/15min: Delefilcon A contact lenses worn bilaterally for 16 waking hours (1 day) in Period 1, followed by 15 minutes in Period 2. A fresh pair of lenses was dispensed for Period 2.
- 15min/16hr: Delefilcon A contact lenses worn bilaterally for 15 minutes in Period 1, follwed by 16 waking hours (1 day) in Period 2. A fresh pair of lenses was dispensed for Period 2.
Period: Period 1, First Wear
Arm/Group | 16hr/15min | 15min/16hr
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0
Period: Period 2, Second Wear
Arm/Group | 16hr/15min | 15min/16hr
Started | 7 | 8
Completed | 7 | 7
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized participants.
Groups:
- Overall: Delefilcon A contact lenses worn during Period 1 and Period 2
Arm/Group | Overall
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (10.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Average Coefficient of Friction (CF) at 16 Hours Compared to Unworn
Description: Worn contact lenses were removed from the participant's eye. The CF was calculated and compared to the CF for unworn contact lenses. A lower CF may indicate higher contact lens lubricity. The ex-vivo lubricity was carried out on one lens (one eye) only.
Time Frame: Day 1 (for each period), 16 hours
Population: This analysis population includes all participants who completed the study.
Measure: Mean (Standard Deviation); unit: unitless
Groups:
- 16 Hours: Delefilcon A contact lenses worn for 16 hours in Period 1 or 2
- Unworn: Unworn delefilcon A contact lenses removed from the commercial packaging and soaked overnight in phosphate buffered saline
Arm/Group | 16 Hours | Unworn
Number analyzed (Participants) | 14 | 14
unitless | 0.0394 (0.0015) | 0.0396 (0.0027)

2. Secondary Outcome: Average Coefficient of Friction at 15 Minutes
Description: Worn contact lenses were removed from the participant's eye and the CF was calculated. A lower CF may indicate higher contact lens lubricity. The ex-vivo lubricity was carried out on one lens (one eye) only.
Time Frame: Day 1 (for each period), 15 minutes
Population: This analysis population includes all participants who completed the study.
Measure: Mean (Standard Deviation); unit: unitless
Groups:
- 15 Minutes: Delefilcon A contact lenses worn for 15 minutes during Period 1 or 2
Arm/Group | 15 Minutes
Number analyzed (Participants) | 14
unitless | 0.0392 (0.0017)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (March 2014 - April 2014). This analysis population includes all participants exposed to the investigational product, based on treatment-specific exposure.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the medical device. AEs were obtained as solicited comments from the study participants and as observations by the Investigator.
Groups:
- DAILIES TOTAL1: Delefilcon A contact lenses worn during Period 1 and Period 2
Arm/Group | DAILIES TOTAL1
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 2/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DAILIES TOTAL1 (N=15)
Corneal infiltrates (Eye disorders) | 1
Ocular discomfort (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes